CLINICAL TRIAL: NCT01533792
Title: Effect of Non-surgical Periodontal Treatment on Pregnant Women With Periodontitis: a Randomized Clinical Trial
Brief Title: Effect of Non-surgical Periodontal Treatment
Acronym: EONSPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Maranhão (Other)
Responsible Party: Principal Investigator, Danielli Maria Zucateli Feitosa, MsC, Universidade Federal do Maranhão
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFMA-2011-DANI
Record Dates: First submitted 2012-01-28; First posted 2012-02-15 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Periodontal Diseases; Adverse Effects
Keywords: Treatment; pregnant women; periodontitis; dental scaling; dental plaque
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Dental Plaque | interventions — Dental Scaling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supra/subgingival therapy (Experimental): The experimental group received supra and subgingival scaling associated with oral hygiene orientation (OHO)
  Interventions: Procedure: Supra/subgingival scaling using periodontal curette scraping; Procedure: Supra and subgingival scaling
- Control group (Active Comparator): Control group received only supragingival scaling with OHO too.
  Interventions: Procedure: Supra/subgingival scaling using periodontal curette scraping; Procedure: Supra and subgingival scaling

INTERVENTIONS:
Procedure: Supra/subgingival scaling using periodontal curette scraping — The experimental group received supra and subgingival therapy with periodontal curettes
Procedure: Supra and subgingival scaling — The experimental group received supra and subgingival scaling.

SUMMARY:
Objective: The objective of this research was to compare the effect of a single session supragingival scaling in a group of pregnant women with periodontal disease with a group that received supra and subgingival scaling.

Methods: The investigators included 34 pregnant women between 15 and 43 who had at least 4 teeth with probing depth ≥ 4 mm or clinical attachment loss ≥ 3 mm, with bleeding on probing in the same place. Women were divided into two groups, the group 1 received supra and subgingival scaling associated with oral hygiene orientation (OHO) and the group 2 received only supragingival scaling with OHO too.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 15 and 43 who had at least 4 teeth with probing depth ≥ 4 mm or clinical attachment loss ≥ 3 mm, with bleeding on probing in the same place.

Exclusion Criteria:

* Patients with systemic disease or who used medications that interfere in the etiological factors of periodontal disease in the last six months, who wore braces and / or prosthetic devices, and women smokers who did not complete treatment.

Ages: 15 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Effect of non-surgical periodontal treatment in pregnancy with periodontal disease | 30 days
  A single calibrated examiner performed clinical examination in pregnant women participating in the measurement of parameters: probing depth, clinical attachment level, hyperplasia, recession, bleeding, presence of plaque and tooth mobility on a standardized form.
  Quantitative parameters were evaluated at six sites per tooth: mesio/medium/ distobuccal and mesio/medium/distolingual through millimeter periodontal probe-type Williams. The bleeding and the presence of plaque in dichotomous variables were measured: present and absent. All patients received oral hygiene orientation (OHO).
Effect of non-surgical periodontal treatment in pregnancy with periodontitis | Assess periodontal disease at times: initial (when pregnancy arrived) and final (30 days after periodontal therapy).
  The patients were randomly divided by lottery into two groups. The group 1, termed SUPRA/SUB received OHO, supra and subgingival scraping and the group 2: SUPRA supragingival scraping and OHO. In both groups, the scaling procedure was performed using periodontal curettes type Mc Call 13-14 and 17-18 (DUFLEX) in one session.
  Within 30 days after the initial session scraping clinical parameters were reevaluated, and now, according to every need, the patients were submitted to the supra and subgingival therapy. Noting that full dental care was provided to participants.